CLINICAL TRIAL: NCT04688892
Title: Immediate Effects of Dynamic Cupping on Median Nerve's Mechanosensitivity, Measured by the Upper Limb Neurodynamic Test 1 (ULNT1) in Healthy Participants: A Randomized Controlled Trial
Brief Title: Immediate Effects of Dynamic Cupping on Median Nerve's Mechanosensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Fernando Pessoa (Other)
Responsible Party: Principal Investigator, Ricardo Cardoso, Clinical Professor, University Fernando Pessoa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FISIO-1-28102019
Record Dates: First submitted 2020-12-03; First posted 2020-12-30 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Healthy
MeSH Terms: interventions — Cupping Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): The type of cupping therapy will be dry-cupping with moving-cupping (dynamic cupping therapy). The participants will remain in the supine position on a massage table (Posturarte® Olympic), without inclination. Cupping therapy will be performed with a plastic suction cup (5.08 cm in diameter) (K.S. Choi Corp®) and with a pistol for dosing pumps (K.S. Choi Corp®). Prior to the cupping therapy, a small amount of massage cream (ATL®) will be applied throughout the median nerve pathway in order to facilitate the sliding of the suction cup. The cupping therapy will performed with the suction cup sliding with a slow rhythm, insufflation of the suction cup with two pumps for 5 minutes along the median nerve path.
  Interventions: Device: Cupping
- Control Group (No Intervention): The participants will remain at rest in a supine position on a massage table (Posturarte® Olympic) without inclination for 5 minutes.

INTERVENTIONS:
Device: Cupping — dynamic cupping
  Arms: Intervention Group

SUMMARY:
The purpose oh this study is to verify the immediate effects of dynamic cupping on median nerve's mechanosensitivity, measured by the upper limb neurodynamic test 1 (ULNT1) in healthy participants.

DETAILED DESCRIPTION:
After completing the socio-demographic and clinical questionnaire, the participants will be randomly assigned into two designated groups, the Intervention Group (IG; n = 30) (dynamic cupping therapy throughout the median nerve course) and the Control Group (CG; n = 30) (remained at rest for 5 minutes), using the software www.graphpad.com/quickcals.

ELIGIBILITY:
Inclusion Criteria:

• Healthy university students of both genders with normal mobility of the joints of the upper quadrant of the body.

Exclusion Criteria:

* Deformities in the upper quadrant region of the body;
* Complaints in this region in the last 6 months;
* Surgical procedures or musculoskeletal, cardiac, renal, metabolic, neurological and or oncological pathologies of the upper quadrant that may disturb nerve function;
* Not present any mechanosensitive response to ULNT1;
* Pregnant women;
* Ingestion of non-steroidal anti-inflammatory drugs or consumption of any type of narcotic drugs and participants who have drunk alcohol in the last 12 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
change in elbow extension range of motion | Baseline (M0), Immediately after intervention or control (M1).
  Data will be collected in two moments: baseline (M0) and after the application of cupping for intervention group or after a resting period for control group (M1).
  The M0 will consist in performing the ULNT1 on the dominant upper limb for each participant. The participants will remain in a supine position on a massage table with the body aligned, exposing the test forearm for the placement of the smartphone through an armband. The head and cervical spine will be stabilized at the maximum comfortable lateral inclination using a foam pillow. The ULNT1 sequence used was: (1) maximum contralateral cervical inclination; (2) arm at 90º of shoulder abduction preventing scapular elevation; (3) 90º of external rotation of the shoulder and elbow flexion at 90º (defined as the initial position or 0º of range of motion under test); (4) supination of the forearm; (5) wrist and fingers extension; and (6) elbow extension.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Cardoso, PhD, Principal Investigator — Fernando Pessoa University
Locations (1):
- Ricardo Cardoso, Porto, Portugal